CLINICAL TRIAL: NCT01301963
Title: Comparison of Plerixafor and G-CSF Versus G-CSF Alone for Stem Cell Mobilization in Patients With Multiple Myeloma Previously Treated With Lenalidomide
Brief Title: Filgrastim With or Without Plerixafor in Treating Patients With Multiple Myeloma Previously Treated With Lenalidomide
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CASE3A10; NCI-2011-00186 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-07

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — plerixafor; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive G-CSF SC QD on days 1-4.
  Interventions: Biological: filgrastim
- Arm II (Experimental): Patients receive G-CSF SC QD on days 1-4 and plerixafor SC QD on days 4-8.
  Interventions: Drug: plerixafor; Biological: filgrastim

INTERVENTIONS:
Drug: plerixafor — Given SC
  Other Names: AMD 3100; Mozobil
  Arms: Arm II
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen

SUMMARY:
This clinical trial studies filgrastim (G-CSF) with or without plerixafor in treating patients with multiple myeloma (MM) previously treated with lenalidomide. Giving colony-stimulating factors, such as G-CSF, and plerixafor helps stem cells move from the patient's bone marrow to the blood so they can be collected and stored

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Ability to reach target collection of 5 x 10^6 CD34+ cells/Kg with =< 2 days of leukaphereses using one of two mobilization regimens.

SECONDARY OBJECTIVES:

I. Percentage of patients achieving target goal CD34+ cell dose (as above) in =< 5 days of leukaphereses.

II. Compare collections between different mobilization regimens in those patients who are crossed over from one mobilization regimen to the other.

III. Compare days of apheresis, need for hospitalization during mobilization, and need for remobilization between mobilizing groups.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive G-CSF subcutaneously (SC) once daily (QD) on days 1-8.

ARM II: Patients receive G-CSF SC QD on days 1-7 and plerixafor SC QD on days 4-7.

After completion of study treatment, patients are followed up at 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM by International Myeloma Working Group Criteria
* In first or second complete or partial remission or stable refractory but not actively progressing myeloma according to the classifications provided by The Center for International Blood & Marrow Transplant Research
* Received at least 2 cycles of lenalidomide therapy
* Patients with MM scheduled to undergo stem cell harvest for possible allogeneic stem cell transplant (ASCT)
* At least 2 weeks since last exposure to lenalidomide
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Prior to the start of mobilization:

  * white blood cell count >/= 2.5 x 10^9/L
  * absolute neutrophil count >/= 1.2 x 10^9/L
  * platelet count >/=100 x 10^9/L
  * creatinine clearance >/= 30mL/minute
* If childbearing potential, must either agree to complete abstinence from heterosexual intercourse or effective means of contraception during stem cell mobilization; female patients will undergo pregnancy test prior to stem cell mobilization therapy

Exclusion Criteria:

* Had prior autologous or allogeneic transplantation
* Received pegfilgrastim within 3 weeks or G-CSF within 14 days of first dose of G-CSF for mobilization
* Failed previous hematopoietic stem cell collections or collection attempts
* Received radiation therapy to the pelvic area
* Received lenalidomide within 2 weeks of first dose of G-CSF for mobilization
* Had received experimental therapy within 4 weeks of enrolling in study
* Current or prior history of other malignancies, excluding basal cell carcinoma of the skin

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hien Duong, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Hillard Lazarus, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Control: Patients receive G-CSF SC QD on days 1-4.
  filgrastim: Given SC
- Arm II: Experimental: Patients receive G-CSF SC QD on days 1-4 and plerixafor SC QD on days 4-8.
  plerixafor: Given SC
  filgrastim: Given SC
Period: Overall Study
Arm/Group | Arm I: Control | Arm II: Experimental
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.40 (4.16) | 56.25 (8.18) | 53.00 (6.15)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Ability to Reach Target Collection of 5 x 10^6 CD34+ Cells/kg
Time Frame: In =< 2 days of leukaphereses
Population: due to low enrollment (10% of anticipated participants), no analysis is being done on data collected in this study
Arm/Group | Arm I: Control | Arm II: Experimental
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Patients Achieving Target Goal CD34+ Cells Dose
Time Frame: In =< 5 days of leukaphereses
Population: Due to low enrollment (10% of anticipated participants), no analysis is being done on data collected in this study
Arm/Group | Arm I: Control | Arm II: Experimental
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Compare Hematopoietic Stem Cells/kg Collections Between Different Mobilization Regimens in Those Patients Who Are Crossed Over From One Mobilization Regimen to the Other
Description: Patients will be randomized to receive either G-CSF or Plerixafor with G-CSF. All patients will undergo at least 2 days of leukopheresis. Cells/kg between these 2 arms will be compared. For those patients that do not reach the target goal will undergo a wash-out period and cross over to the other study arm.
Time Frame: By day 1
Reporting Status: Not Posted

4. Secondary Outcome: Compare Days of Apheresis Between Mobilization Groups
Description: Using the Wilcoxon Rand Sum Test
Time Frame: Day 1
Reporting Status: Not Posted

5. Secondary Outcome: Compare Need for Hospitalization During Mobilization Between Mobilization Groups
Time Frame: Day 1
Reporting Status: Not Posted

6. Secondary Outcome: Compare Need for Remobilization Between Mobilization Groups
Description: Using the Chi-square test or Fisher's exact test, as appropriate.
Time Frame: Day 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arm I: Control | Arm II: Experimental
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes